CLINICAL TRIAL: NCT05798000
Title: Effect of WHO Surgical Safety Checklist and Anaesthesia Equipment Checklist on Patients Outcomes in Low-resource Settings.
Brief Title: Effect of WHO Surgical Safety Checklist and Anesthesia Equipment Checklist on Patients Outcomes in Low-resource Settings.
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, Assistant professor at the Department of OF SURGERY, ANESTHESIOLOGY AND INTENSIVE THERAPY OF POSTGRADUATE EDUCATION, Bogomolets National Medical University
Other Study IDs: GF230548
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Safety Issues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: The control group without WHO and equipment checklist used
- Study: Other group, where WHO safety check-list and equipment check-list were implemented

SUMMARY:
The study to investigate the effectiveness and the current perception of safety checklists in Ukrainian hospitals.

DETAILED DESCRIPTION:
A prospective multicenter study was conducted in 6 large Ukrainian hospitals: Kyiv City Clinical Hospitals #1, University Clinic of the Bogomolets National Medical University, Kyiv City Maternity Hospital #5, National Cancer Institute, Shalimov National Institute of Surgery and Transplantology, Saint Martin Hospital in Mukachevo. Institutions were selected among those, where surgical department administration was willing to implement the Safe Surgery Saves Lives campaign recommendations, but has not yet formally introduced the WHO Safe Surgery Checklist. On each study site, 1 or 2 operating rooms were designated for data collection. All surgical procedures observed by the data collectors in those operating rooms were included. The study was conducted in two phases: control period, lasting from February 1, 2022 until August 1, 2022, followed by a week-long educational period during which the WHO Surgical Safety Checklist and the Anesthesia Equipment Checklist were used but no data were collected. The intervention period began on August 8, 2022 and lasted until December 31, 2022. Hospital administration and members of all surgical teams were informed of the nature of the study and the proper checklist use method by the involved anesthesiologists, who were previously instructed by the primary investigators. WHO Surgical Safety Checklists and the Anesthesia Equipment Checklists were provided in the designated operating rooms. Both checklists were translated into Ukrainian. The requirement for written informed consent from the patient was waived by the ethical committee of Bogomolets National Medical University. The study design was approved by the ethics committee of the Bogomolets National Medical University (protocol #148, 07.09.2021).

ELIGIBILITY:
Inclusion Criteria:

* medical institutions with surgical departments

Exclusion Criteria:

* medical institutions without surgical departments

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Institutions, where surgical department administration was willing to implement the Safe Surgery Saves Lives campaign recommendations but has not yet formally introduced the WHO Safe Surgery Checklist.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Recorded critical incidents during the procedure | 24 hours
  Recorded critical incidents during the procedure (hypotension, hypertension etc.)
Mortality | 28 days
  Postoperative mortality during 28 days after surgery

SECONDARY OUTCOMES:
Postoperative complications | 1 months
  Postoperative complications (bleeding, surgical infection etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Kateryna Bielka, PhD, Study Director — Bogomolets National Medical University
Locations (1):
- Bogomolets NMU, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwendimann R, Blatter C, Luthy M, Mohr G, Girard T, Batzer S, Davis E, Hoffmann H. Adherence to the WHO surgical safety checklist: an observational study in a Swiss academic center. Patient Saf Surg. 2019 Mar 12;13:14. doi: 10.1186/s13037-019-0194-4. eCollection 2019. PMID 30918531
- [Background] Sendlhofer G, Mosbacher N, Karina L, Kober B, Jantscher L, Berghold A, Pregartner G, Brunner G, Kamolz LP. Implementation of a surgical safety checklist: interventions to optimize the process and hints to increase compliance. PLoS One. 2015 Feb 6;10(2):e0116926. doi: 10.1371/journal.pone.0116926. eCollection 2015. PMID 25658317
- [Background] Bergs J, Hellings J, Cleemput I, Zurel O, De Troyer V, Van Hiel M, Demeere JL, Claeys D, Vandijck D. Systematic review and meta-analysis of the effect of the World Health Organization surgical safety checklist on postoperative complications. Br J Surg. 2014 Feb;101(3):150-8. doi: 10.1002/bjs.9381. PMID 24469615